CLINICAL TRIAL: NCT03505671
Title: Acupuncture for Chemotherapy-Induced Peripheral Neuropathy Among Breast Cancer Patients
Brief Title: Acupuncture in Reducing Chemotherapy-Induced Peripheral Neuropathy in Participants With Stage I-III Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00049061; NCI-2018-00586 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 97118 (Other: Wake Forest University Health Sciences); P30CA012197 (NIH)
Record Dates: First submitted 2018-04-12; First posted 2018-04-23 (Actual); Results first posted 2022-05-11 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Grade 1 Peripheral Motor Neuropathy, CTCAE; Grade 1 Peripheral Sensory Neuropathy, CTCAE; Grade 2 Peripheral Motor Neuropathy, CTCAE; Grade 2 Peripheral Sensory Neuropathy, CTCAE; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: interventions — Acupuncture Therapy; Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (acupuncture) (Experimental): Participants undergo 8 45-minute acupuncture treatments over 10 weeks.
  Interventions: Procedure: Acupuncture Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group 2 (usual care) (Active Comparator): Participants receive usual care.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Acupuncture Therapy — Undergo acupuncture therapy
  Other Names: Acupuncture
  Arms: Group 1 (acupuncture)
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Group 2 (usual care)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
The goal of this study is to obtain preliminary evidence of the effect of 8 acupuncture treatments over 10 weeks in breast and GI cancer patients who are currently receiving or recently completed active neurotoxic chemotherapy and have clinically documented grade 1 or 2 neuropathy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To obtain preliminary evidence of the clinical effects of acupuncture compared to usual care on the change in sensory neuropathic pain as measured by the European Organization of Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-Chemotherapy-Induced Peripheral Neuropathy (CIPN) 20 item (20) sensory subscale.

SECONDARY OBJECTIVES:

I. Change in the motor and autonomic neuropathic pain subscores on the EORTC QLQ-CIPN20.

II. Change in patient-reported assessment of numbness and tingling using the 2-item Patient-Reported Outcomes (PRO)-Common Terminology Criteria for Adverse Events (CTCAE) measure.

III. Preventing the escalation of CIPN from grade 1 or 2 to a higher grade. IV. Amount and intensity of planned chemotherapy relative to completed chemotherapy.

V. Effect on sensory and motor nerve function via nerve conduction studies (NCS) (e.g. conduction velocity, latency, and amplitude).

VI. Effect on peripheral nerve swelling via nerve ultrasound (e.g. cross sectional area, CSA).

EXPLORATORY OBJECTIVES:

I. To obtain preliminary evidence on phenotypic differences between African-American and non African-American (A-A) (i.e., white, Asian, etc.) with regard to presentation of CIPN as well as response to the intervention.

II. To obtain preliminary evidence of the effect of acupuncture on intraepidermal nerve fiber density (IENF) via skin biopsy.

III. To examine the associations among the peripheral nerve assessment measures (nerve conduction, peripheral nerve ultrasound, skin biopsy) and of the peripheral nerve assessment measures with the patient reported outcomes (EORTC QLQ-CIN20, PRO-CTCAE) at baseline, week 12, and for the change from baseline to week 12.

IV. To examine the association between expectations of the effectiveness of acupuncture to reduce peripheral neuropathy and baseline, 12 week, and change in patient-reported outcomes on the EORTC QLQ-CIPN20 and PRO-CTCAE.

OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP 1: Participants undergo 8 45-minute acupuncture treatments over 10 weeks.

GROUP 2: Participants receive usual care.

After completion of study treatment, participants are followed up at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Breast and GI cancer stage I-III
* Currently receiving or recently completed neurotoxic chemotherapy (either adjuvant or neoadjuvant). Currently is defined as including up until when the next cycle would be delivered, that is if the patient is getting chemotherapy every week, this would include a week after their last treatment; if the patient is getting treatment every 2 weeks, this would include 2 weeks after their last treatment; if the patient is getting treatment every 3 weeks, this would include 3 weeks after their last treatment, etc. Recently completed is defined as 6 weeks after this time period. For example, if a patient was getting chemotherapy every week, this would include seven weeks after their last treatment; if the patient was getting treatment every 2 weeks, this would include 8 weeks after their last treatment; if the patient were getting treatment every 3 weeks, this would include 9 weeks after their last treatment, etc.
* Clinical symptoms of peripheral neuropathy of grade 1 or grade 2 as measured by the National Cancer Institute (NCI)-CTCAE
* Ability and willingness to understand and sign an informed consent

Exclusion Criteria:

* Self-reported or documented history of UNRESOLVED pre-existing peripheral neuropathy due to diabetes, human immunodeficiency virus (HIV), or other conditions.
* Unable to provide medical history.
* Male patients.
* Pregnant.
* Unwilling to receive acupuncture or unable to travel for treatments.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Avis, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 (Acupuncture) | Group 2 (Usual Care)
Started | 11 | 12
Completed | 8 | 11
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Acupuncture) | Group 2 (Usual Care) | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (10.6) | 56.8 (12.5) | 56.5 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 12 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 9 | 8 | 17
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in the Sensory Neuropathic Pain Score as Measured by the European Organization of Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-Chemotherapy-Induced Peripheral Neuropathy (CIPN) 20 Item (20)
Description: Will estimate means and standard deviations by group for the EORTC QLQ-CIPN20 sensory subscale, the correlation between the two measures, and the within-person change. To estimate effect size, we will use an analysis of covariance (ANCOVA) model at week 12, which will include the group and the baseline value. Using a 4-point Likert scale (1 = "not at all," 2 = "a little," 3 = "quite a bit," and 4 = "very much"), individuals indicate the degree to which they have experienced sensory, motor, and autonomic symptoms during the past week. Sensory raw scale scores range from 1 to 36, motor raw scale scores range from 1 to 32, and autonomic raw scale scores range from 1 to 12 for men and 1-8 for women (erectile function item is excluded) [13]. All scale scores are linearly converted to a 0-100 scale, with higher scores indicating more symptom burden.
Time Frame: Baseline up to week 12
Population: Number of participants analyzed may differ due to participants being lost to follow up or withdrawing from intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (Acupuncture) | Group 2 (Usual Care)
Number analyzed (Participants) | 10 | 12
score on a scale
  Baseline | 16.7 (3.7) | 17.5 (3.0)
  Week 12: number analyzed (Participants) | 9 | 11
  Week 12 | 13.7 (2.7) | 14.8 (5.2)
  Week 12 - Baseline (Change): number analyzed (Participants) | 9 | 11
  Week 12 - Baseline (Change) | -2.9 (4.2) | -2.5 (5.8)
Statistical Analysis 1: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.61, ANCOVA
Statistical Analysis 2: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; Correlation Coefficient = 0.15 — Correlation between EORTC Sensory Subscale baseline and 12 weeks (overall, N=20)
Statistical Analysis 3: Comparison: Group 1 (Acupuncture); Test type: Other; Correlation coefficient = 0.25 — Correlation between EORTC Sensory Subscale baseline and 12 weeks (intervention, N=9)
Statistical Analysis 4: Comparison: Group 2 (Usual Care); Test type: Other; Correlation coefficient = 0.09 — Correlation between EORTC Sensory Subscale baseline and 12 weeks (Usual Care, N=11)

2. Secondary Outcome: Change in Motor and Autonomic Pain Subscores on the EORTC QLQ-CIPN20
Description: Means and standard deviations will be computed at baseline and week 12 by group, and for the change in the measures, and will also estimate the correlation between the measures at the two time points, and fit ANCOVA models for each outcome. Using a 4-point Likert scale (1 = "not at all," 2 = "a little," 3 = "quite a bit," and 4 = "very much"), individuals indicate the degree to which they have experienced sensory, motor, and autonomic symptoms during the past week. Sensory raw scale scores range from 1 to 36, motor raw scale scores range from 1 to 32, and autonomic raw scale scores range from 1 to 12 for men and 1-8 for women (erectile function item is excluded). All scale scores are linearly converted to a 0-100 scale, with higher scores indicating more symptom burden.
Time Frame: Baseline up to week 12
Population: Number of participants analyzed may differ due to participants being lost to follow up or withdrawing from intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (Acupuncture) | Group 2 (Usual Care)
Number analyzed (Participants) | 10 | 12
score on a scale
  Baseline EORTC Subscale | 11.1 (3.2) | 11.3 (2.1)
  Week 12 EORTC Subscale: number analyzed (Participants) | 9 | 11
  Week 12 EORTC Subscale | 11.0 (1.8) | 11.1 (3.3)
  Week 12 - Baseline (Change) EORTC Subscale: number analyzed (Participants) | 9 | 11
  Week 12 - Baseline (Change) EORTC Subscale | 0.1 (2.2) | -0.1 (2.7)
  Baseline EORTC Autonomic Subscale | 2.7 (0.9) | 2.8 (0.8)
  Week 12 - EORTC Autonomic Subscale: number analyzed (Participants) | 9 | 11
  Week 12 - EORTC Autonomic Subscale | 2.4 (0.7) | 2.3 (0.5)
  Week 12 - Baseline EORTC Autonomic Subscale: number analyzed (Participants) | 9 | 11
  Week 12 - Baseline EORTC Autonomic Subscale | -0.3 (1.1) | -0.5 (0.9)
Statistical Analysis 1: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.91, ANCOVA — P value for the motor subscale
Statistical Analysis 2: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.55, ANCOVA — P value for autonomic subscale

3. Secondary Outcome: Change in Patient-Reported Outcomes (PRO)-Common Terminology Criteria for Adverse Events (CTCAE) Measure of Numbness and Tingling
Description: Means and standard deviations will be computed at baseline and week 12 by group, and for the change in the measures, and will also estimate the correlation between the measures at the two time points, and fit ANCOVA models for each outcome. The CTCAE measure of CIPN will be assessed using frequencies of grade by time point (baseline, week 12), as well as whether the grade of CIPN increased, decreased or remained stable. A Fisher's Exact test will be used to compare the groups at each time point and for the change during the study period.
Time Frame: Baseline up to week 12
Population: Number of participants analyzed may differ due to participants being lost to follow up or withdrawing from intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Acupuncture) | Group 2 (Usual Care)
Number analyzed (Participants) | 10 | 12
Participants
  Baseline - Numbness or Tingling Severity (None 1) | 4 | 2
  Baseline - Numbness or Tingling Severity (Mild 2) | 3 | 8
  Baseline - Numbness or Tingling Severity (Moderate 3) | 2 | 1
  Baseline - Numbness or Tingling Severity (Severe 4) | 1 | 1
  Baseline - Numbness or Tingling Severity (Very severe 5) | 0 | 0
  Week 12 - Numbness or Tingling Severity (None 1): number analyzed (Participants) | 9 | 11
  Week 12 - Numbness or Tingling Severity (None 1) | 1 | 2
  Week 12 - Numbness or Tingling Severity (Mild 2): number analyzed (Participants) | 9 | 11
  Week 12 - Numbness or Tingling Severity (Mild 2) | 6 | 4
  Week 12 - Numbness or Tingling Severity (Moderate 3): number analyzed (Participants) | 9 | 11
  Week 12 - Numbness or Tingling Severity (Moderate 3) | 2 | 3
  Week 12 - Numbness or Tingling Severity (Severe 4): number analyzed (Participants) | 9 | 11
  Week 12 - Numbness or Tingling Severity (Severe 4) | 0 | 0
  Week 12 - Numbness or Tingling Severity (Very severe 5): number analyzed (Participants) | 9 | 11
  Week 12 - Numbness or Tingling Severity (Very severe 5) | 0 | 0
  Baseline - Numbness or Tingling Interference - Not at all (1) | 4 | 1
  Baseline - Numbness or Tingling Interference - A little bit (2) | 2 | 7
  Baseline - Numbness or Tingling Interference - Somewhat (3) | 2 | 2
  Baseline - Numbness or Tingling Interference -Quite a bit (4) | 2 | 2
  Baseline - Numbness or Tingling Interference - Very much (5) | 0 | 0
  Week 12 - Numbness or Tingling Interference - Not at all (1): number analyzed (Participants) | 9 | 11
  Week 12 - Numbness or Tingling Interference - Not at all (1) | 3 | 7
  Week 12 - Numbness or Tingling Interference - A little bit (2): number analyzed (Participants) | 9 | 11
  Week 12 - Numbness or Tingling Interference - A little bit (2) | 5 | 1
  Week 12 - Numbness or Tingling Interference - Somewhat (3): number analyzed (Participants) | 9 | 11
  Week 12 - Numbness or Tingling Interference - Somewhat (3) | 1 | 3
  Week 12 - Numbness or Tingling Interference - Quite a bit (4): number analyzed (Participants) | 9 | 11
  Week 12 - Numbness or Tingling Interference - Quite a bit (4) | 0 | 0
  Week 12 - Numbness or Tingling Interference - Very much (5): number analyzed (Participants) | 9 | 11
  Week 12 - Numbness or Tingling Interference - Very much (5) | 0 | 0
  Week 12 - Baseline (Change) Numbness or Tingling Severity (Decreased, less than or equal to -1): number analyzed (Participants) | 9 | 11
  Week 12 - Baseline (Change) Numbness or Tingling Severity (Decreased, less than or equal to -1) | 5 | 7
  Week 12 - Baseline (Change) Numbness or Tingling Severity - Same (0): number analyzed (Participants) | 9 | 11
  Week 12 - Baseline (Change) Numbness or Tingling Severity - Same (0) | 3 | 1
  Week 12 - Baseline (Change) Numbness or Tingling Severity (Increased, >/= 1): number analyzed (Participants) | 9 | 11
  Week 12 - Baseline (Change) Numbness or Tingling Severity (Increased, >/= 1) | 1 | 3
  Week 12 - Baseline (Change) Numbness or Tingling Interference - (Decreased, </= -1): number analyzed (Participants) | 9 | 11
  Week 12 - Baseline (Change) Numbness or Tingling Interference - (Decreased, </= -1) | 3 | 7
  Week 12 - Baseline (Change) Numbness or Tingling Interference - (Same - 0): number analyzed (Participants) | 9 | 11
  Week 12 - Baseline (Change) Numbness or Tingling Interference - (Same - 0) | 5 | 3
  Week 12 - Baseline (Change) Numbness or Tingling Interference - (Increased, >/= -1): number analyzed (Participants) | 9 | 11
  Week 12 - Baseline (Change) Numbness or Tingling Interference - (Increased, >/= -1) | 1 | 1
Statistical Analysis 1: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.41, Fisher Exact — P value for baseline numbness or tingling severity data
Statistical Analysis 2: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.22, Fisher Exact — P value for baseline numbness or tingling interference data
Statistical Analysis 3: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.58, Fisher Exact — Week 12 p value for numbness or tingling severity data
Statistical Analysis 4: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.12, Fisher Exact — P value for Week 12 numbness or tingling interference data
Statistical Analysis 5: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.57, Fisher Exact — Week 12 - Baseline p value for numbness or tingling severity data
Statistical Analysis 6: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.55, Fisher Exact — Week 12 - Baseline p value for numbness or tingling interference

4. Secondary Outcome: CIPN as Measured by National Cancer Institute (NCI)-CTCAE 5.0 Grades 1-3 Numbness or Tingling
Description: The CTCAE measure of CIPN will be assessed using frequencies of grade by time point (baseline, week 12), as well as whether the grade of CIPN increased, decreased or remained stable. A Fisher's Exact test will be used to compare the groups at each time point and for the change during the study period.
Time Frame: Up to week 12
Population: Number of participants analyzed may differ due to participants being lost to follow up or withdrawing from intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Acupuncture) | Group 2 (Usual Care)
Number analyzed (Participants) | 11 | 12
Participants
  Baseline - Grade 1 Numbness or Tingling | 10 | 10
  Baseline - Grade 2 Numbness or Tingling | 1 | 2
  Baseline - Grade 3 Numbness or Tingling | 0 | 0
  Week 12 - Grade 1 Numbness or Tingling: number analyzed (Participants) | 8 | 11
  Week 12 - Grade 1 Numbness or Tingling | 7 | 9
  Week 12 Grade 2 Numbness or Tingling: number analyzed (Participants) | 8 | 11
  Week 12 Grade 2 Numbness or Tingling | 1 | 1
  Week 12 Grade 3 Numbness or Tingling: number analyzed (Participants) | 8 | 11
  Week 12 Grade 3 Numbness or Tingling | 0 | 1
  Week 12 - Baseline Numbness or Tingling Severity Decreased (</= 1): number analyzed (Participants) | 8 | 11
  Week 12 - Baseline Numbness or Tingling Severity Decreased (</= 1) | 0 | 0
  Week 12 - Baseline Numbness or Tingling Severity Same (0): number analyzed (Participants) | 8 | 11
  Week 12 - Baseline Numbness or Tingling Severity Same (0) | 7 | 9
  Week 12 - Baseline Numbness or Tingling Severity Increased (>/= 1): number analyzed (Participants) | 8 | 11
  Week 12 - Baseline Numbness or Tingling Severity Increased (>/= 1) | 1 | 2
Statistical Analysis 1: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.99, Fisher Exact — P value for baseline numbness or tingling severity Grade 1-3
Statistical Analysis 2: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.99, Fisher Exact — P value for 12 weeks numbness or tingling severity Grade 1-3
Statistical Analysis 3: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.99, Fisher Exact — P value for week 12 - baseline change in numbness or tingling severity

5. Secondary Outcome: Number of Participants With Standard Chemotherapy Dose or Decreased Due to Peripheral Neuropathy
Description: Means and standard deviations will be computed at baseline and week 12 by group, and will also estimate the correlation between the measures at the two time points
Time Frame: Up to week 12
Population: Number of participants analyzed may differ due to participants being lost to follow up or withdrawing from intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Acupuncture) | Group 2 (Usual Care)
Number analyzed (Participants) | 9 | 10
Participants
  Chemotherapy dose standard | 6 | 7
  Chemotherapy dose decreased due to chemotherapy induced peripheral neuropathy | 3 | 3
Statistical Analysis 1: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.99, Fisher Exact

6. Secondary Outcome: Number of Cycles of Completed Chemotherapy
Description: Means and standard deviations will be computed at baseline and week 12 by group, and will also estimate the correlation between the measures at the two time points, and fit ANCOVA models for each outcome.
Time Frame: Up to week 12
Population: Number of participants analyzed may differ due to participants being lost to follow up or withdrawing from intervention.
Measure: Mean (Standard Deviation); unit: cycles
Arm/Group | Group 1 (Acupuncture) | Group 2 (Usual Care)
Number analyzed (Participants) | 9 | 11
cycles | 4.4 (0.7) | 4.2 (1.0)
Statistical Analysis 1: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.69, t-test, 2 sided

7. Secondary Outcome: Cross Sectional Area (CSA) of Peripheral Nerves as Determined by Ultrasound (Sural and Median)
Description: as for outcome 6
Time Frame: Up to week 12
Population: Number of participants analyzed may differ due to participants being lost to follow up or withdrawing from intervention. Treatment ended early for 2 participants in the intervention group, discontinued the intervention
Measure: Mean (Standard Deviation); unit: meters squared
Arm/Group | Group 1 (Acupuncture) | Group 2 (Usual Care)
Number analyzed (Participants) | 9 | 12
meters squared
  Baseline - Cross sectional area - sural | 3.1 (1.5) | 2.8 (0.7)
  Baseline - Cross sectional area - median | 14.2 (6.3) | 12.7 (3.3)
  Week 12 - Cross sectional area - sural: number analyzed (Participants) | 9 | 11
  Week 12 - Cross sectional area - sural | 3.0 (1.3) | 3.0 (1.2)
  Week 12 - Cross sectional area - median: number analyzed (Participants) | 9 | 11
  Week 12 - Cross sectional area - median | 14.6 (7.5) | 11.9 (2.8)
  Week 12 - Baseline - Cross sectional area - sural (Change): number analyzed (Participants) | 7 | 11
  Week 12 - Baseline - Cross sectional area - sural (Change) | -0.4 (1.0) | 0.1 (1.3)
  Week 12 - Baseline - Cross sectional area - median (Change): number analyzed (Participants) | 7 | 11
  Week 12 - Baseline - Cross sectional area - median (Change) | 0.1 (1.5) | -1.0 (2.0)
Statistical Analysis 1: Comparison: Group 1 (Acupuncture); Test type: Other; p = 0.46, ANCOVA — P value for cross sectional area sural data
Statistical Analysis 2: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.22, ANCOVA — P value for cross sectional area for median data

8. Secondary Outcome: Amplitude of Nerve Response Derived From Nerve Conduction Studies (NCS) (Sural, Tibial, and Median)
Description: Means and standard deviations will be computed at baseline and week 12 by group, and will also estimate the correlation between the measures at the two time points, and fit ANCOVA models for each outcome. Nerve conduction studies measure impairment of electrical function in large peripheral nerves and measures amplitude and latency of neuronal signaling. Ranging from 0.1 μm to 20 μm. Reduction in the amplitude indicates axonal damage.
Time Frame: Up to week 12
Population: Number of participants analyzed may differ due to participants being lost to follow up or withdrawing from intervention.
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Group 1 (Acupuncture) | Group 2 (Usual Care)
Number analyzed (Participants) | 9 | 12
micrometers
  Baseline - Amplitude (sural) | 9.5 (5.0) | 9.5 (7.6)
  Week 12 - Amplitude (sural) | 8.8 (3.6) | 10.9 (7.8)
  Week 12 - Baseline Amplitude (sural) | -1.5 (4.6) | 0.7 (1.8)
  Baseline - Amplitude - Tibial, ankle | 13.3 (5.6) | 11.0 (3.8)
  Week 12 - Amplitude - Tibial, ankle: number analyzed (Participants) | 8 | 10
  Week 12 - Amplitude - Tibial, ankle | 12.4 (5.2) | 11.5 (3.5)
  Week 12 - Baseline - Amplitude - Tibial, ankle (Change): number analyzed (Participants) | 8 | 12
  Week 12 - Baseline - Amplitude - Tibial, ankle (Change) | -1.5 (1.9) | -0.2 (1.7)
  Baseline - Amplitude - Tibial, pop fossa | 8.5 (5.2) | 7.8 (3.7)
  Week 12 - Amplitude - Tibial, pop fossa: number analyzed (Participants) | 8 | 12
  Week 12 - Amplitude - Tibial, pop fossa | 10.0 (4.4) | 7.9 (3.0)
  Week 12 - Baseline - Amplitude - Tibial, pop fossa (Change): number analyzed (Participants) | 8 | 12
  Week 12 - Baseline - Amplitude - Tibial, pop fossa (Change) | 1.0 (3.4) | -0.8 (1.9)
  Baseline - Amplitude - median, wrist | 9.6 (3.6) | 10.3 (2.8)
  Week 12 - Amplitude - median, wrist: number analyzed (Participants) | 8 | 12
  Week 12 - Amplitude - median, wrist | 10.1 (4.4) | 11.2 (2.7)
  Week 12 - Baseline - Amplitude - median, wrist (Change): number analyzed (Participants) | 8 | 12
  Week 12 - Baseline - Amplitude - median, wrist (Change) | 0.1 (3.3) | 0.4 (2.4)
  Baseline - Amplitude - median, elbow: number analyzed (Participants) | 8 | 12
  Baseline - Amplitude - median, elbow | 9.3 (3.7) | 10.0 (2.8)
  Week 12 - Amplitude - median, elbow: number analyzed (Participants) | 8 | 12
  Week 12 - Amplitude - median, elbow | 9.3 (4.0) | 10.8 (2.7)
  Week 12 - Baseline Amplitude - median, elbow (Change): number analyzed (Participants) | 7 | 12
  Week 12 - Baseline Amplitude - median, elbow (Change) | -0.3 (3.1) | 0.5 (2.3)
Statistical Analysis 1: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.20, ANCOVA — P value for amplitude - sural data
Statistical Analysis 2: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.28, ANCOVA — P value for amplitude - tibial, ankle
Statistical Analysis 3: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.13, ANCOVA — P value for amplitude tibial, pop fossa
Statistical Analysis 4: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.71, ANCOVA — P value for amplitude median, wrist
Statistical Analysis 5: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.46, ANCOVA — P value for amplitude, median, elbow

9. Secondary Outcome: Distal Latency of Nerve Response Derived From NCS (Sural, Tibial, and Median)
Description: as for outcome 6
Time Frame: Up to week 12
Population: Number of participants analyzed may differ due to participants being lost to follow up or withdrawing from intervention.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Group 1 (Acupuncture) | Group 2 (Usual Care)
Number analyzed (Participants) | 9 | 12
milliseconds
  Baseline - Latency Sural: number analyzed (Participants) | 9 | 10
  Baseline - Latency Sural | 3.4 (0.6) | 3.4 (0.6)
  Week 12 - Latency Sural: number analyzed (Participants) | 9 | 10
  Week 12 - Latency Sural | 3.4 (0.6) | 3.3 (0.6)
  Week 12 -Baseline - Latency Sural (Change): number analyzed (Participants) | 9 | 10
  Week 12 -Baseline - Latency Sural (Change) | 0.0 (0.7) | 0.0 (0.3)
  Baseline - Latency tibial, ankle | 3.6 (0.3) | 4.0 (0.5)
  Week 12 - Latency tibial, ankle: number analyzed (Participants) | 8 | 10
  Week 12 - Latency tibial, ankle | 3.6 (0.5) | 3.8 (0.6)
  Week 12 - Baseline Latency tibial, ankle (Change): number analyzed (Participants) | 8 | 10
  Week 12 - Baseline Latency tibial, ankle (Change) | -0.1 (0.8) | -0.2 (0.4)
  Baseline - Latency tibial, pop | 11.5 (1.0) | 11.7 (1.2)
  Week 12 - Latency tibial, pop: number analyzed (Participants) | 8 | 10
  Week 12 - Latency tibial, pop | 11.2 (1.1) | 11.5 (1.2)
  Week 12 - Baseline Latency tibial, pop: number analyzed (Participants) | 8 | 10
  Week 12 - Baseline Latency tibial, pop | -0.2 (0.6) | 0.1 (0.4)
  Baseline - Latency median wrist | 4.0 (1.1) | 3.7 (0.5)
  Week 12 - Latency median wrist: number analyzed (Participants) | 8 | 10
  Week 12 - Latency median wrist | 4.4 (1.9) | 3.7 (0.5)
  Week 12 - Baseline Latency median wrist (Change: number analyzed (Participants) | 8 | 10
  Week 12 - Baseline Latency median wrist (Change | 0.5 (1.0) | -0.1 (0.4)
  Baseline - Latency median elbow | 7.8 (1.5) | 7.5 (0.7)
  Week 12 - Latency median elbow: number analyzed (Participants) | 8 | 10
  Week 12 - Latency median elbow | 8.2 (2.5) | 7.5 (0.7)
  Week 12 - Baseline - Latency median elbow (Change): number analyzed (Participants) | 8 | 10
  Week 12 - Baseline - Latency median elbow (Change) | 0.4 (1.2) | 0.0 (0.6)
Statistical Analysis 1: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.81, ANCOVA — P value for latency sural data
Statistical Analysis 2: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.76, ANCOVA — P value for latency tibial, ankle data
Statistical Analysis 3: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.24, ANCOVA — P value for latency tibial, pop fossa
Statistical Analysis 4: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.20, ANCOVA — P value for latency median wrist data
Statistical Analysis 5: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.51, ANCOVA — P value for latency median elbow data

10. Secondary Outcome: Conduction Velocity of Nerve Response Derived From NCS (Sural, Tibial, and Median)
Description: as for outcome 6
Time Frame: Up to week 12
Population: Number of participants analyzed may differ due to participants being lost to follow up or withdrawing from intervention. Two participants in the intervention group discontinued the intervention/treatment earlier than the anticipated 12 weeks time frame.
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Group 1 (Acupuncture) | Group 2 (Usual Care)
Number analyzed (Participants) | 9 | 12
meters per second
  Baseline - Velocity Sural: number analyzed (Participants) | 9 | 10
  Baseline - Velocity Sural | 51.1 (3.0) | 45.9 (3.8)
  Week 12 - Velocity Sural: number analyzed (Participants) | 8 | 9
  Week 12 - Velocity Sural | 50.5 (5.6) | 48.7 (4.2)
  Week 12 - Baseline Velocity Sural (Change): number analyzed (Participants) | 8 | 9
  Week 12 - Baseline Velocity Sural (Change) | -1.0 (6.6) | 2.2 (3.6)
  Baseline - Velocity Tibial | 49.1 (3.3) | 50.3 (5.1)
  Week 12 - Velocity Tibial: number analyzed (Participants) | 8 | 10
  Week 12 - Velocity Tibial | 51.1 (5.6) | 49.4 (5.4)
  Week 12 - Baseline - Velocity Tibial (Change): number analyzed (Participants) | 8 | 10
  Week 12 - Baseline - Velocity Tibial (Change) | 2.1 (4.3) | -2.0 (2.3)
  Baseline - Velocity Median: number analyzed (Participants) | 8 | 12
  Baseline - Velocity Median | 55.5 (3.7) | 54.2 (4.1)
  12 Weeks - Velocity Median: number analyzed (Participants) | 8 | 10
  12 Weeks - Velocity Median | 55.3 (5.9) | 55.5 (2.8)
  Week 12 - Baseline - Velocity Median (Change): number analyzed (Participants) | 7 | 10
  Week 12 - Baseline - Velocity Median (Change) | -0.6 (5.3) | 0.1 (2.9)
Statistical Analysis 1: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.98, ANCOVA — P value for velocity sural data
Statistical Analysis 2: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.03, ANCOVA — P value for velocity tibial data
Statistical Analysis 3: Comparison: Group 1 (Acupuncture) vs Group 2 (Usual Care); Test type: Other; p = 0.81, ANCOVA — P value for velocity median data

11. Secondary Outcome: Nerve Fiber Density in the Skin
Description: as for outcome 6
Time Frame: Up to week 12
Population: Number of participants analyzed may differ due to participants being lost to follow up or withdrawing from intervention.
Measure: Mean (Standard Deviation); unit: fibers per millimeter
Arm/Group | Group 1 (Acupuncture) | Group 2 (Usual Care)
Number analyzed (Participants) | 4 | 7
fibers per millimeter
  Baseline - Nerve fiber density, distal leg | 7.8 (3.2) | 8.3 (3.3)
  Week 12 - Nerve fiber density, distal leg: number analyzed (Participants) | 3 | 2
  Week 12 - Nerve fiber density, distal leg | 3.5 (0.7) | 4.3 (1.7)
  Week 12 - Baseline - Nerve fiber density, distal leg: number analyzed (Participants) | 3 | 2
  Week 12 - Baseline - Nerve fiber density, distal leg | -5.1 (2.8) | -4.5 (3.0)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Group 1 (Acupuncture) | Group 2 (Usual Care)
All-Cause Mortality (participants affected / at risk) | 0/11 | 1/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (Acupuncture) (N=11) | Group 2 (Usual Care) (N=12)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/71/NCT03505671/Prot_SAP_001.pdf
  • Informed Consent Form (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/71/NCT03505671/ICF_002.pdf